CLINICAL TRIAL: NCT00921830
Title: A Single-dose, Randomised, Crossover Study to Compare the Rate and Extent of Absorption of Three Formulations of Ibuprofen in Healthy, Fasting Male and Female Volunteers
Brief Title: Pharmacokinetics of 3 Formulations of Ibuprofen Suppositories
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SCO2203
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: ibuprofen; healthy volunteers; bioavailability; pharmacokinetics; suppository
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibuprofen (Experimental): ibuprofen
  Interventions: Drug: ibuprofen

INTERVENTIONS:
Drug: ibuprofen — Each subject will receive single doses of (i) ibuprofen 50 mg suppository (ii) ibuprofen 200 mg suppository and (iii) ibuprofen 200 mg tablet in 3 separate dosing periods. Doses will be administered after an overnight fast.
  Other Names: MOTRIN®

SUMMARY:
The purpose of this study is to compare the pharmacokinetic and bioavailability characteristics of two test formulations of ibuprofen for rectal administration with the profile of a marketed reference formulation of ibuprofen 200 mg (for oral administration).

DETAILED DESCRIPTION:
Ibuprofen is a widely used analgesic and antipyretic in adults and children. Two ibuprofen suppository formulations have been developed for pediatric use to facilitate dosing in younger age groups. This is a single-dose, balanced, randomised, three-period crossover study in healthy male and female adult volunteers. Each volunteer will receive a single dose of 50 mg ibuprofen as a suppository, a single dose of 200 mg ibuprofen as a suppository and a single oral dose of 200 mg ibuprofen (tablet). There will be 14 blood samples taken over 12 hours in each study period. Concentrations in plasma of ibuprofen and its S and R enantiomers will be measured using a validated chromatographic method. Standard pharmacokinetic parameters will be obtained and bioavailability on the basis of rate and extent of drug absorption will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged between 18 and 55 years
* BMI < 27 kg/m2
* Non-smokers, or smokers of less than 10 cigarettes per day
* Clinically normal vital signs
* Clinically normal medical history
* Clinically normal findings on physical examination
* Clinically normal findings for haematology and clinical chemistry of blood and urine or showing clinically insignificant deviations only
* Screening results for drug abuse (taken within 14 days of study start) must be negative for opiates, cannabinoids, amphetamines, methamphetamine, benzodiazepines and cocaine
* HIV and Hepatitis B and C tests, taken within previous 14 days of study start, must be negative
* Appropriate use of an effective method of contraception (female volunteers only). Use of the oral contraceptive pill is permitted
* Ability to comprehend and communicate effectively with the Investigator and staff
* Ability to give written informed consent
* Electrocardiogram recording (12-lead) within the normal range

Exclusion Criteria:

* History of peptic ulcer or gastrointestinal bleeding
* Resting heart rate outside the range 50 - 90 beats per minute or exhibiting any clinically significant degree of heart block
* Resting, seated blood pressure less than 100/60 (90/50 for females) or greater than 140/90 mmHg
* Clinically significant electrolyte imbalance
* Evidence of clinically significant cardiovascular, haematological, hepatic, gastrointestinal, renal, respiratory, neurological, or psychiatric disease
* History of medication with any psycho-pharmacologically active agents within the last five years (other than occasional night sedatives)
* Gastric bleeding or history of allergies to NSAIDs
* History of psychiatric illness or clinical treatment for psychiatric illness within the last five years
* History of epilepsy
* History of significant drug or drug related hypersensitivity/intolerance or food allergies
* Illness within 14 days prior to start of study
* Hospitalisation within the previous 3 months for major surgery or significant medical illness (at the discretion of the Investigator)
* Mental handicap as defined by clinical evaluation
* Tobacco smoking of more than 10 cigarettes per day
* Participation in a clinical drug study in which blood was taken within 16 weeks prior to the start of the study
* Donation of blood or plasma within previous 90 days
* Participation in a clinical trial in the previous 12 months in which a volume of blood exceeding 500 ml was donated
* Any indication of current or previous abuse of alcohol, solvents or drugs
* Treatment with a full or regular course of medication during the 28 days prior to the start of the study
* Use of alcohol on study days or within 24 hours prior to commencement of each study period
* Intake of grapefruit products within 7 days prior to study commencement
* Intake of methylxanthine-containing beverages within 24 hours prior to each study period
* Intake of quantities of methylxanthine or alcohol-containing beverages which, in the opinion of the Investigator are abnormal (habitually taking more than 5 cups or glasses of tea, coffee, cola, chocolate etc per day or habitually taking more than 20g alcohol/day)
* Taking medication (prescription or proprietary) within 14 days prior to the study start. Paracetamol is allowed up to 72 hours prior to either study period. The oral contraceptive pill is allowed.
* Failure to use adequate contraceptive measures; positive pregnancy test (female volunteers only)
* Lactating/breastfeeding (female volunteers only)
* Diet, which in the opinion of the Investigator, deviates from a normal diet (e.g. vegans)
* Not able/not willing to give informed consent
* Not able to be contacted in case of emergency.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2004-04; Primary Completion 2004-07 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, including AUC0-t and AUC0-∞ | 14 samples over 12 hours in each period

SECONDARY OUTCOMES:
Pharmacokinetic parameters, including Cmax, tmax, t1/2 and Terminal Elimination Rate Constant | 14 samples over 12 hours in each period

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Cottrell, Study Director — McNeil UK
Locations (1):
- Shandon Clinic, Cork, Co. Cork, Ireland